CLINICAL TRIAL: NCT03264599
Title: Measurement of the Fetal Occiput-spine Angle During the First Stage of Labor as Predictor of the Maternal and Fetal Outcome of Labor
Brief Title: Measurement of the Fetal Occiput-spine Angle During the First Stage of Labor as Predictor of the Outcome of Labor
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Professor, Cairo University
Other Study IDs: 12
Record Dates: First submitted 2017-08-25; First posted 2017-08-29 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Vaginal Delivery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- occiput-spine angle > or = 126: 2D trans abdominal ultrasound was done during the first stage of labor. If fetal position is occiput anterior and fetal presentation is vertex, two dimensional sagittal picture of the fetal head and upper spine was acquired and stored in the ultrasound machine. On this image, the offline measurement of the angle formed by a line tangential to the occipital bone and a line tangential to the first vertebral body of the cervical spine (occiput-spine angle > or = 126) will be performed to quantify the degree of fetal head flexion in respect to the trunk
  Interventions: Device: transabdominal ultrasound
- occiput-spine angle<126: 2D trans abdominal ultrasound was done during the first stage of labor. If fetal position is occiput anterior and fetal presentation is vertex, two dimensional sagittal picture of the fetal head and upper spine was acquired and stored in the ultrasound machine. On this image, the offline measurement of the angle formed by a line tangential to the occipital bone and a line tangential to the first vertebral body of the cervical spine (occiput-spine angle < 126) will be performed to quantify the degree of fetal head flexion in respect to the trunk
  Interventions: Device: transabdominal ultrasound

INTERVENTIONS:
Device: transabdominal ultrasound — 2D trans abdominal ultrasound was done during the first stage of labor. If fetal position is occiput anterior and fetal presentation is vertex, two dimensional sagittal picture of the fetal head and upper spine was acquired and stored in the ultrasound machine. On this image, the offline measurement of the angle formed by a line tangential to the occipital bone and a line tangential to the first vertebral body of the cervical spine (occiput-spine angle) will be performed to quantify the degree of fetal head flexion in respect to the trunk

SUMMARY:
2D trans abdominal ultrasound was done during the first stage of labor. If fetal position is occiput anterior and fetal presentation is vertex, two dimensional sagittal picture of the fetal head and upper spine was acquired and stored in the ultrasound machine. On this image, the offline measurement of the angle formed by a line tangential to the occipital bone and a line tangential to the first vertebral body of the cervical spine (occiput-spine angle) will be performed to quantify the degree of fetal head flexion in respect to the trunk

DETAILED DESCRIPTION:
2D trans abdominal ultrasound was done during the first stage of labor. If fetal position is occiput anterior and fetal presentation is vertex, two dimensional sagittal picture of the fetal head and upper spine was acquired and stored in the ultrasound machine. On this image, the offline measurement of the angle formed by a line tangential to the occipital bone and a line tangential to the first vertebral body of the cervical spine (occiput-spine angle) will be performed to quantify the degree of fetal head flexion in respect to the trunk.

The sonographer was not involved in the patient's care and the managing obstetrician was blinded to the ultrasound findings and the occiput-spine angle. For each patient of the study group, the progress of labor using a partogram ( cervical dilation ,effacement ,consistency, position and station ) and the mode of delivery were assessed retrospectively.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 & 35 years old.
2. BMI is less than 30
3. The gestational age between 37- 42 weeks. (calculated by LMP or 1st trimesteric U/S)
4. Singleton pregnancy.
5. History of one vaginal delivery.
6. Occiputo anterior position.
7. Active phase of first stage of labor.

Exclusion Criteria:

1. Age (below18 or above 35).
2. Primigravida.
3. Occiputo posterior position.
4. Indications of cesarean section like malpresentations , macrosomia , placenta previa, previous cesarean section .
5. Multiple gestation.
6. Medical disorders like hypertension, DM, liver or renal diseases

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: a total of 400 women with gestational age 37 weeks or more and history of one vaginal delivery at least
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2016-07-11 (Actual); Primary Completion 2017-07-21 (Actual); Study Completion 2017-08-20 (Actual)

PRIMARY OUTCOMES:
vaginal delivery | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — kasr Alainy medical school
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided